CLINICAL TRIAL: NCT01417754
Title: Volume and Circulation Changes of The Breast in 3D Ultrasound During Toremifene Versus Nonmedicated Menstrual Cycle
Brief Title: Changes in Breast 3D Ultrasound Measurements Using Toremifene
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Satakunta Central Hospital (Other)
Collaborators: Tampere University Hospital (Other); Tampere University (Other)
Responsible Party: Principal Investigator, SINIKKA OKSA, MD, principal investigator, Satakunta Central Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Tore3D
Record Dates: First submitted 2011-07-28; First posted 2011-08-16 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Circulatory; Change
Keywords: toremifene
MeSH Terms: interventions — Toremifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Toremifene (Other)
  Interventions: Drug: Toremifene

INTERVENTIONS:
Drug: Toremifene — 20mg toremifene per day in tablet form starting from the cycle day 15 and continued to premenstrual period. Medication using about 10 days per volunteer
  Other Names: trade name Fareston

SUMMARY:
To investigate if there are detectable changes in volume and circulation in breasts of healthy volunteers using toremifene 20 mg in luteal phase of the menstruation cycle versus nonmedicated cycle.

DETAILED DESCRIPTION:
20 women were participated to this trial.

ELIGIBILITY:
Inclusion Criteria:

* age 25-45 healthy person
* regular menstrual cycles
* safe contraception(for example sterilization or condom)

Exclusion Criteria:

* gynecological or other type of cancer
* hormonal contraception
* pregnancy

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
circulation changes of the breast | cycle day 23 to 26

CONTACTS AND LOCATIONS:
Overall Officials: Sinikka Oksa, MD, Principal Investigator — Satakunta Central Hospital; Johanna Mäenpää, professor, Study Director — Tampere University Hospital
Locations (1):
- Porin Lääkäritalo, Pori, Finland